CLINICAL TRIAL: NCT05207683
Title: Pulmonary Hypertension in Patients Attending Sohag University Hospital: A Focus on The Etiology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Abdo Saad, Assistant lecturer of chest diseases and tuberculosis sohag university hospitals, Sohag University
Other Study IDs: Soh-Med-21-12-20
Record Dates: First submitted 2021-12-29; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Patients With Pulmonary Hypertension
MeSH Terms: interventions — X-Rays; Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with pulmonary hypertension: patients who are more than 18 years old , diagnosed with pulmonary hypertension by echocardiography
  Interventions: Other: echocardiography

INTERVENTIONS:
Other: echocardiography — All the patients will be subjected to thorough medical history and clinical examination and the results of the previous investigations will be collected aiming for reaching the diagnosis of the etiology of pulmonary hypertension. ct pulmonary angiography and then right heart catheterization will be done in case of undiagnosed etiology.
  Other Names: electrocardiogram; chest X ray; high resolution Ct chest; spirometry; arterial blood gases; abdominal ultrasound; CT pulmonary angiography; serological tests e.g Anti nuclear antibodies, anti double stranded DNA antibodies...; right heart catheterization

SUMMARY:
Assessment of pulmonary hypertension in patients attending Sohag university hospital ( in out patient clinic or in patient) focusing on the etiology of pulmonary hypertension

ELIGIBILITY:
Inclusion Criteria:

* patients who are 18 years old or more
* patients with pulmonary hypertension diagnosed with echocardiography

Exclusion Criteria:

* patient who are less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pulmonary hypertension patients attending Sohag university hospital (either admitted in the hospital or attending the out patient clinics)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Detection of the causes of pulmonary hypertension in patients attending Sohag university hospital | one year
  We will diagnose the cause of pulmonary hypertension in each participant. This will be done by following the diagnostic algorithm of European Society of Cardiology/ European Respiratory Society (ESC/ERS) 2015 guidelines (e.g. we will exclude that pulmonary hypertension is secondary to pulmonary disease by performing adequate assessment of the patient medical history and clinical examination, performing chest x-ray and or high resolution CT chest, spirometry...), so we will know the pattern of pulmonary hypertension etiology in patients attending of Sohag university hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prins KW, Thenappan T. World Health Organization Group I Pulmonary Hypertension: Epidemiology and Pathophysiology. Cardiol Clin. 2016 Aug;34(3):363-74. doi: 10.1016/j.ccl.2016.04.001. PMID 27443134
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] Simonneau G, Montani D, Celermajer DS, Denton CP, Gatzoulis MA, Krowka M, Williams PG, Souza R. Haemodynamic definitions and updated clinical classification of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801913. doi: 10.1183/13993003.01913-2018. Print 2019 Jan. PMID 30545968